CLINICAL TRIAL: NCT05246657
Title: EUS-guided Entero-biliary Anastomosis as Fistulas for Therapeutic Access in Benign Biliary Obstructions Not Accessible by ERCP
Brief Title: EUS-guided Entero-biliary Anastomosis for Therapeutic Access in Benign Biliary Obstructions
Acronym: ATENHEA
Status: Recruiting | Type: Observational
Sponsor: Hospital del Rio Hortega (Other)
Responsible Party: Principal Investigator, Marina de Benito Sanz, Principal Investigator, Hospital del Rio Hortega
Other Study IDs: ATENHEA
Record Dates: First submitted 2022-02-04; First posted 2022-02-18 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- intervention: EUS-guided Entero-biliary Anastomosis
  Interventions: Procedure: EUS-guided Entero-biliary Anastomosis

INTERVENTIONS:
Procedure: EUS-guided Entero-biliary Anastomosis — EUS-guided Entero-biliary Anastomosis

SUMMARY:
Background: Transpapillary EUS-BD (rendezvous/antegrade) is gaining acceptance in BBO. The potential of transmural EUS-BD (hepaticogastrostomy/choledochoduodenostomy) in complex BBO warrants study.

Aims: To assess feasibility and efficacy of TEA using transmural covered self-expandable metal-stents (cSEMS) to provide interval biliary drainage and create TAF for biliary endotherapy under cholangioscopy or fluoroscopy in BBO not amenable to ERCP.

DETAILED DESCRIPTION:
3.1 Design

Prospective multicenter case series

3.1 Design

Prospective multicenter case series

3.2 Study population

The study population includes patients with benign biliary obstruction in whom a temporary enterobiliary anastomosis is considered by transmural stent deployment. All consecutive patients who meet inclusion criteria and do not present exclusion criteria identified in the endoscopy units of the Río Hortega University Hospital in Valladolid will be invited to participate.

3.4. Intervention

Patients who meet the inclusion criteria and do not present any exclusion criteria (preendoscopic) will be invited to participate in the study. The informed consent will be completed in accordance with Law 41/2002 on patient autonomy without altering the relationship with your doctor or causing any damage to your treatment.

1. Pre-endoscopic management

   A clinical assessment of the patient will be carried out (history, physical examination)
2. Endoscopic procedure:

   All patients will receive antibiotic prophylaxis before the procedure according to the currentguidelines. Endoscopic interventions will be performed under sedation by expert endoscopists in tertiary centers with or without the participation of residents.

   -The EUS-guided enterobiliary anastomosis technique is performed as follows: a standard therapeutic channel echoendoscope (GF-UCT 180; Olympus Europa) is inserted into the stomach or jejunum to allow endosonographic view of left liver lobe. Intrahepatic ducts of adequate caliber are identified avoiding the intervening vessels identified by Doppler. In the case of EUS-guided choledocochoduodenostomy (EUS-CD), the echoendoscope is passed into the duodenum to visualize the common bile duct and its proper caliber. A 19-gauge needle (Expect; Boston Scientific, Marlborough, Mass) preloaded with water-soluble contrast material is used to puncture in the selected duct through the liver, and entry is confirmed by injection of contrast. The needle is cleaned with saline and a 0.025-inch, 450-cm-long hydrophilic-tipped guidewire (VisiGlide; Olympus Spain) is passed antegrade toward the biliary tree. The needle is withdrawn and, in case of intrahepatic puncture, the tract is ballon-dilated(CRE controlled radial expansion balloon dilator; Boston Scientific) directly over the guide wire. Balloon dilation begins from within the left intrahepatic duct and continues sequentially to the tip of the endoscope and through the gastric or intestinal wall. the tract was dilated with a biliary dilation balloon (CRE controlled radial expansion balloon dilator; Boston Scientific ) directly over the guide wire. Sequential balloon dilation fromthe left intrahepatic duct into the tip of the endoscope,is performed through the gastric or intestinal wall. the tract was dilated with a biliary dilation balloon (CRE controlled radial expansion balloon dilator; Boston Scientific) directly over the guide wire. Balloon dilatation begins from within the left intrahepatic duct and continues sequentially to the tip of the endoscope and through the gastric or intestinal wall.

   Subsequently, a stent is deployed under radiological and endoscopic ultrasound view, , creating the enterobiliary anastomosis. The type and size of the stent, as well as the option of using anchoring methods or not, will be chosen at the discretion of the endoscopist and will be collected in the database.
   * After performing the anastomosis, one or more therapeutic sessions will be carried out through the stent or, removing it, through the bare fistula. The first of these sessions can be carried out on the same day as the fistula or on a deferred basis. The techniques carried out on each of the sessions will depend on the initial indication.
   * Once the useful life of the enterobiliary fistula has ended, that is, when the endoscopist decides that the therapeutic sessions have ended, either by achieving clinical success or by opting for surgical or percutaneous rescue, the stentwill be removed endoscopically, registering in the CRD the technique used for it.
3. Follow-up:

It will be carried out through contact with your doctors/responsible nursing staff after 24 hours, and through in-personor telephone visits depending on availability and the patient's clinical situation 7 days after performing the enterobiliary fistula, 24 hours after each one of the endoscopic sessions and at 24h, 30 days and at 3 and 6 months (+/- 5 days) after removal of the stent Esta parte no la entiendo muy bien.

During the visits, the clinical situation, blood tests with complete blood count and liver function parameters and possible unidentified complications will be collected. The visit at 24 hours is part of normal clinical practice, since the patient is usually kept under observation until the day after the procedure, to confirm the absence of immediate complications.

3.5 Sample size

The studies available on this type of procedure have a small number of cases, given that they are highly specialized techniques, which are performed only in reference hospitals by expert personnel. We do not have studies that evaluate the variability between operators in this type of procedure, therefore it is difficult to estimate a minimum sample size. Taking into account the number of procedures performed in the participating centers, our goal is to include a minimum of 50 procedures.

3.6 Data collection

All the variables concerning the characteristics of the procedure, type of stent and the complications that occurred will be collected in each center. The variables concerning follow-up will be collected centrally, through in-personor telephone visits with the responsible physicians, which will be carried out 24 hours after each endoscopic session, and through face-to-face or telephone visits depending on availability and the clonic ?? situation of the patient. patient 7 days after making the fistula and 30 days and 3 and 6 months after removal of the prosthesis.

3.7 Data handling

The CRF data will be entered by the principal investigator or collaborating investigators anonymously, encrypted and dissociated from the clinical information by means of a patient identification code (ID), in an online database. The responsible physician, who is also a researcher, will define an ID for each patient, whose relationship with the clinical history will only be accessible by him, with its custody in a file protected by a personal password. The data entered in the database will be anonymous and the database will be protected with a password to which only researchers will have access.

With regard to the application of the Organic Law on Data Protection 15/1999 and Royal Decree 1720/2007 that develops it, it should be noted that the protocol defined in the project aimed at epidemiological analysis determines that the files will record information completely anonymized. A file will be kept with the information compiled for the development of the project within the framework defined in the Security Document of the maximum level of the Río Hortega University Hospital, whose responsibility is the Management of this organization. this document is public, of obligatory knowledge and available on the Intranet of the Río Hortega University Hospital. The levels of security, access and availability will be those defined in this document.

3.8 Statistical analysis

Categorical variables will be described as percentages. Continuous with normal distribution as mean and standard deviation. Continuous variables with non-normal distributions will be described as medians and interquartile range (the range may also be offered). The analysis will be performed using Stata (StataCorp. 2016. College Station, Texas).

4. ETHICAL ASPECTS

4.1 Benefit-risk assessment for research subjects

The benefit we seek is to assess the efficacy and safety profile of enterobiliary anastomosis as a therapeutic access fistula in benign biliary obstructions. We consider that participating in the study does not imply a significant increase in the usual risks in these patients, given that it is a purely observational project. Performing an endoscopic ultrasound-guided bilioenteroanastomosis presents risks similar to those assumed during any advanced therapeutic endoscopy (perforation, gastrointestinal bleeding, migration of the stent).

As technical aspects of the study, the stents are those usually used for the creation of this type of anastomosis, being an indication included in the current technical data sheet of the product.

4.2. Data Confidentiality

The study data will initially be dissociated from the identity of the participant, by means of an ID, by the responsible physician. The relationship between the ID and the identity of the participant will be kept by the research doctors in a file protected with a personal password. The data will be entered into the database encrypted with the participant's ID, to maintain their anonymity. The database will be password protected and only accessible by researchers. During the study, strict compliance with Law 3/2018 on the Protection of Personal Data is guaranteed.

ELIGIBILITY:
Inclusion Criteria:

* • Consecutive patients ≥ 18 years old.

  * Benign biliary obstruction.
  * ERCP failed or where ERCP could not be performed due to surgically-altered anatomy

Exclusion Criteria:

* • Refusal to sign the informed consent.

  * Malignant biliary obstruction
  * Coagulopathy (INR>1.5) or trombocytopenia (<50,000 platelets/mm3) uncorrectable.
  * Inability to tolerate the sedation necessary for the examination.
  * Pregnancy or lactation.
  * Unable to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population includes patients with benign biliary obstruction in whom a temporary enterobiliary anastomosis is considered by transmural stent deployment. All consecutive patients who meet inclusion criteria and do not present exclusion criteria identified in the endoscopy units of the Río Hortega University Hospital in Valladolid will be invited to participate.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Clinical success | 1 year
  Change major or equal than 2 mg/dl of total bilirrubine

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Maroto Martin, PI, Principal Investigator — Hospital Rio Hortega
Locations (1):
- Hospital Rio Hortega, Valladolid, Spain

IPD SHARING:
Plan to Share IPD: No